CLINICAL TRIAL: NCT05153525
Title: Continuous Infusion Versus Intermittent Boluses of Cisatracurium in the Early Management of Pediatric Acute Respiratory Distress Syndrome
Brief Title: Continuous Infusion Versus Intermittent Boluses of Cisatracurium in the Early Management of Pediatric ARDS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Khaled Talaat, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34409/1/21
Record Dates: First submitted 2021-09-13; First posted 2021-12-10 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Distress Syndrome, Pediatric; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
Keywords: Cisatracurium; PARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intermittent boluses group (Experimental): Thirty children with ARDS will be managed with intermittent boluses of Cisatracurium (0.1-0.15 mg/kg/dose).
  Interventions: Drug: Intermittent boluses of Cisatracurium
- Intravenous infusion for 24 hours (Experimental): Thirty children with ARDS will be treated with intravenous infusion of Cisatracurium titrated from 1 mic/kg/min till reaching the desired effect for 24 hours.
  Interventions: Drug: Intravenous infusion of Cisatracurium for 24 hours

INTERVENTIONS:
Drug: Intermittent boluses of Cisatracurium — Thirty children with ARDS will be treated with intermittent boluses of Cisatracurium (0.1-0.15 mg/kg/dose).
  Arms: Intermittent boluses group
Drug: Intravenous infusion of Cisatracurium for 24 hours — Thirty children with ARDS will be treated with intravenous infusion of Cisatracurium titrated from 1 mic/kg/min till reaching the desired effect for 24 hours.
  Arms: Intravenous infusion for 24 hours

SUMMARY:
The aim of this work is to compare continuous infusion vs on need intermittent boluses of Cisatracurium in the early management of pediatric acute respiratory distress syndrome

DETAILED DESCRIPTION:
In the pediatric population, Acute respiratory distress syndrome (ARDS) has a high mortality rate of approximately 24%. In addition, there is a lack of high-quality data to guide the use of non-depolarizing neuromuscular blocking agents (NMBAs) in mechanically ventilated children. Hence, there is a need to evaluate its use in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

1. Children with mild, moderate, and severe ARDS diagnosed according to criteria of Pediatric Acute Lung Injury Consensus Conference (PALICC) in 2015.
2. Children of both sexes aged from one month to 18 years.
3. Children diagnosed with ARDS <48 hours before enrollment

Exclusion Criteria:

1. Continuous neuromuscular blockade at enrollment
2. Children on phenytoin and carbamazepine
3. Severe liver cirrhosis
4. High-risk medical illness (Bone marrow transplantation within the last one-year, Diffuse alveolar hemorrhage from vasculitis, Chronic respiratory failure, Burns > 70% total body surface)
5. Previous hypersensitivity or anaphylactic reaction to Cisatracurium
6. Neuromuscular conditions that may potentiate neuromuscular blockade and/or impair effective spontaneous ventilation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-05 (Estimated)

PRIMARY OUTCOMES:
Duration on mechanical ventilation | Up to 10 days
  Time from patient's intubation till extubation

SECONDARY OUTCOMES:
Length of pediatric intensive care unit stay | 28 days
  Time from start of ventilation till discharge from PICU
Length of hospital stay | 28 days
  Time from start of ventilation till discharge from hospital
Pediatric intensive care unit acquired weakness | 28 days
  Manual muscle strength testing (Oxford testing)
Organ failure free days to day 28 | 28 days
  Organ failure according to SOFA scores
Ventilation follow-up | 7 days
  Oxygenation Index/Oxygen saturation index on study days 1, 3, 7
28-day mortality | 28 days
  All children died after mechanical ventilation till day 28
Serum Interleukin-8 assessment | 48 hours
  Assessing serum interleukin 8 on admission and after 48 hours
Mechanical ventilation complications follow-up | 28 days
  Development of pneumothorax during mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Khaled Talaat, PharmD, Principal Investigator — Tanta University
Locations (2):
- Egypt (2):
  - Tanta University Hospitals, Tanta, Gharbia Governorate
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: for one year after completion of the study